CLINICAL TRIAL: NCT06061809
Title: Open-Label, Single-Arm Phase 2 Study of Nogapendekin Alfa Inbakicept, PD-L1 t-haNK, Bevacizumab and Randomized Phase 2B Study of Nogapendekin Alfa Inbakicept, Bevacizumab, and Tumor Treatment Fields With or Without PD-L1 t-haNK in Participants With Recurrent or Progressive Glioblastoma
Brief Title: N-803 and PD-L1 t-haNK Combined With Bevacizumab for Recurrent or Progressive Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.078
Record Dates: First submitted 2023-09-12; First posted 2023-09-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: Progressive Glioblastoma; Recurrent Glioblastoma; N-803; ALT-803; PD-L1 t-haNK; Immunotherapy; Bevacizumab; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Arm (Experimental): Phase 2
  Participants will receive N-803 1 mg subcutaneously (SC), PD-L1 t-haNK (~2 × 10^9 cells/infusion) intravenously (IV), and Bevacizumab (10 mg/kg IV) combination therapy during 28-day cycles on days 1 and 15 of each cycle. Maximum treatment period is 76 weeks, 19 cycles.
  Interventions: Drug: Bevacizumab; Drug: PD-L1 t-haNK; Drug: N-803
- Experiment Treatment Arm A (Experimental): Phase 2B: Participants will be randomized 1:1 to 1 of 2 experimental arms (Arm A or Arm B). Treatment for all enrolled participants will consist of repeated 8-week cycles for a maximum treatment period of up to 80 weeks (10 cycles).
  Experimental Arm (A):
  Every 2 weeks (Days 1, 15, 29, and 43 of an 8-week cycle):
  N-803, 1 mg SC Bevacizumab, 10 mg/kg IV Continuous application (≥ 18 hours/day) to the brain: TTFields, 200 kHz
  Interventions: Drug: Bevacizumab; Drug: N-803; Device: Tumor Treating Fields (TTFields, 200 kHz)
- Experiment Treatment Arm B (Experimental): Participants will be randomized 1:1 to 1 of 2 experimental arms (Arm A or Arm B). Treatment for all enrolled participants will consist of repeated 8-week cycles for a maximum treatment period of up to 80 weeks (10 cycles).
  Every 2 weeks (Days 1, 15, 29, and 43 of an 8-week cycle):
  PD-L1 t-haNK, 2 × 109 cells per infusion IV NAI, 1 mg SC Bevacizumab, 10 mg/kg IV
  Plus - Continuous application (≥ 18 hours/day) to the brain: TTFields, 200 kHz
  Interventions: Drug: Bevacizumab; Drug: PD-L1 t-haNK; Drug: N-803; Device: Tumor Treating Fields (TTFields, 200 kHz)

INTERVENTIONS:
Drug: Bevacizumab — Participants will receive 10mg/kg of Bevacizumab intravenously (IV) on Day 1 and Day 15 of each repeated cycle of treatment.
  Other Names: Avastin
Drug: PD-L1 t-haNK — Participants will receive PD-L1 t-haNK (~2 × 109 cells/infusion) intravenously (IV) on Day 1 and Day 15 of each repeated cycle of treatment.
  Arms: Experiment Treatment Arm B; Single Arm
Drug: N-803 — Participants will receive 1mg subcutaneously (SC) on Day 1 and Day 15 of each repeated cycle of treatment.
  Other Names: ALT-803; Anktiva
Device: Tumor Treating Fields (TTFields, 200 kHz) — TTFields (OPTUNE Gio®), for the treatment of newly diagnosed and/or recurrent GBM, is a portable battery or power supply operated device which produces alternating electrical fields, called tumor treatment fields ("TTFields") within the human body/brain. TTFields are applied to the patient by electrically-insulated surface transducer arrays. TTFields disrupt the rapid cell division exhibited by cancer cells. TTFields is comprised of two main components: (1) an Electric Field Generator and (2) INE Insulated Transducer Arrays (the transducer arrays). Patients carry the device in an over-the-shoulder bag or backpack and receive continuous treatment without changing their daily routine.
  Arms: Experiment Treatment Arm A; Experiment Treatment Arm B

SUMMARY:
This study consists of 2 portions. The phase 2 portion is an open-label, single-arm study to evaluate the safety and efficacy of NAI, PD-L1 t-haNK, and bevacizumab combination therapy in participants with recurrent or progressive GBM. The phase 2B portion is an open-label, randomized study to evaluate the efficacy and safety for the following 2 experimental arms in participants with recurrent or progressive GBM: NAI, bevacizumab, and TTFields combination therapy (Arm A) or NAI, PD-L1 t-haNK, bevacizumab, and TTFields combination therapy (Arm B).

Phase 2 Treatment for all enrolled participants will consist of repeated cycles of 28 days for a maximum treatment period of 76 weeks (19 cycles) as follows: Every 2 weeks (Days 1 and 15 of a 28-day cycle)

Fourteen (14) participants were enrolled in the phase 2 portion of this study as of the date of this v02 protocol. No additional participants will be administered therapy in phase 2.

Phase 2B Participants will be randomized 1:1 to 1 of 2 experimental arms (Arm A or Arm B). Treatment for all enrolled participants will consist of repeated 8-week cycles for a maximum treatment period of up to 80 weeks (10 cycles). Experimental Arm (A): Every 2 weeks (Days 1, 15, 29, and 43 of an 8-week cycle)

Up to twenty (20) participants will be randomized in phase 2B (up to 10 participants/arm.

Duration of Treatment:

Participants will receive study treatment for up to 76 weeks during phase 2 (up to 19 repeated 28-day cycles) and for up to 80 weeks (up to 10 repeated 8-week cycles) during phase 2B or until they report unacceptable toxicity (not corrected with dose reduction), withdraw consent, or if the Investigator feels it is no longer in the participant's best interest to continue treatment. Treatment may also be discontinued if the participant has confirmed PD per iRANO, unless the participant is clinically stable and is considered potentially deriving benefit per Investigator's assessment.

Duration of Follow-up:

Participants who discontinue study treatment should remain in the study for follow-up. Participants should be followed for collection of survival status, posttreatment therapies (phase 2 and phase 2B), and medical history (phase 2B only) every 12 weeks (± 2 weeks) for the first 2 years then yearly thereafter for an additional 3 years. The maximum duration of follow-up is 5 years (260 weeks).

ELIGIBILITY:
Phase 2 Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed glioblastoma in accordance with the 2021 WHO Classification of Tumors of the CNS (WHO CNS5) that has progressed after initial therapy or therapies. The digital image to be provided for confirmation of histology by the Sponsor. Gliosarcoma, small cell GBM or other GBM variants, and molecular GBM are allowed.
4. Progressive or recurrent disease will be confirmed (i.e. contrast enhanced magnetic resonance imaging (MRI) performed within 3 weeks prior to study treatment per RANO criteria or diagnostic biopsy).
5. Previous first line treatment with at least radiotherapy and temozolomide. Subjects must have been off prior treatment at least 28 days prior to initiation of study therapy. Subjects must be at least 90 days from completion of radiation to reduce the risk of pseudoprogression being misdiagnosed as progression, unless the recurrence is a new enhancement on MRI outside the radiation treatment field or progression is confirmed by biopsy.
6. Subjects must have recovered from prior treatment-related toxicities to Grade 2 or less.
7. Life expectancy > 12 weeks.
8. Karnofsky Performance Status ≥ 70.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 6 months after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 6 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.
11. Craniotomy must be adequately healed (at least 28 days between study treatment initiation and surgery).

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drugs used in this study or that would put the subject at high risk for treatment related complications.
2. Prior anticancer treatment of glioblastoma with bevacizumab or other anti-angiogenic treatment.
3. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 8 mg/day dexamethasone), excluding inhaled steroids. Short-term steroid use to prevent intravenous (IV) contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
4. History of surgery in the past 28 days or with surgical wound not healed.
5. History of serious hemorrhage as defined by NCI CTCAE 5.0 grading.
6. Evidence of > Grade 1 CNS hemorrhage on the baseline MRI scan.
7. History of recent hemoptysis.
8. Subjects receiving therapeutic anticoagulation.
9. Subjects with a history or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.
10. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease) requiring any treatment within the last 5 years.
11. History of organ transplant requiring immunosuppression.
12. History of active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
13. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
14. Body weight ≤ 40 kg at screening.
15. Inadequate organ function, evidenced by the following laboratory results:

    1. Absolute neutrophil count (ANC) < 1,000 cells/mm3.
    2. Hemoglobin < 9 g/dL.
    3. Platelet count < 100,000 cells/mm3.
    4. Total bilirubin > 2 × upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
    5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
    6. Alkaline phosphatase (ALP) levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or > 10 × ULN in subjects with bone metastases).
    7. Serum creatinine > 2.0 mg/dL or 177 µmol/L.
    8. Albumin < 3.0 g/dL.

    Note: Each study site should use its institutional Upper Limit of Normal (ULN) to determine eligibility.
16. Clinically significant (ie, active) cardiovascular disease or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
17. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
18. Known hypersensitivity to any component of the study medication(s).
19. Participation in an investigational drug study or receiving any investigational treatment within 28 days prior to study treatment. No wash out is necessary for subjects previously receiving Tumor treating field (TTF); TTF will be allowed to continue at the discretion of the Investigator. FDA-authorized drugs for the prevention and treatment of COVID-19 are permitted.
20. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
21. Concurrent participation in any interventional clinical trial.
22. Pregnant and nursing women.

Phase 2B Inclusion Criteria

1. Age ≥ 22 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed GBM in accordance with the 2021 WHO CNS5 (grade 4 Glioma, IDH-wildtype) that has progressed after initial therapy or therapies (prior surgical resection if feasible, plus radiotherapy with concurrent and/or adjuvant temozolomide), limited to first-line progression. A second surgical resection is allowed but not required. Gliosarcoma, small cell GBM or other GBM variants, and molecular GBM are allowed.
4. Progressive or recurrent disease will be confirmed (ie, contrast enhanced magnetic resonance imaging [MRI] performed within 4 weeks prior to study treatment per RANO v02 criteria or diagnostic biopsy), or progression that does not meet RANO v02 criteria if the disease progression is otherwise obvious in the opinion of the Investigator and is discussed with the Medical Monitor. Participants must be a minimum of 3 months from the completion of radiotherapy to distinguish true progression from pseudoprogression.
5. Previous first-line treatment with at least radiotherapy and temozolomide.
6. Have received and recovered from standard treatments. At least 4 weeks since any cytotoxic chemotherapy (eg, temozolomide/nitrosoureas), 28 days since any investigational agent, and 6 to 12 weeks since radiation before starting study drug(s).
7. Willingness to use TTFields device. Both experimental arms require wearing the TTFields device ≥ 18 hours a day. Participants must be willing to shave their head twice a week and use the TTFields device as instructed. They should have no scalp condition or implanted device that contraindicates TTFields use (eg, no non-MRI-safe metal in the skull, ventricular peritoneal shunt is generally okay, but no active scalp infections or wounds).
8. Life expectancy ≥ 12 weeks.
9. ECOG performance status of 0 to 2.
10. Have recovered from prior treatment-related toxicities to grade 2 or less.
11. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
12. Agreement to practice highly effective contraception for female participants of childbearing potential and nonsterile males. Female participants of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Female participants of childbearing potential must have a negative pregnancy test and adhere to using a highly effective method of contraception (eg, tubal ligation, approved hormonal contraceptive, or an intrauterine device [IUD]) prior to screening and agree to continue its use during the study or be surgically sterilized (eg, hysterectomy) while on study and for 7 months post last dose of study drug. Male participants must agree to use barrier methods of birth control while on study and for 7 months post last dose of study drug.
13. Craniotomy must be adequately healed (at least 28 days between study treatment initiation and surgery).

Exclusion Criteria:

1. Received any further therapy beyond initial first-line therapy other than surgical resection.
2. Prior therapy with bevacizumab for GBM.
3. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drugs used in this study or that would put the participant at high risk for treatment-related complications.
4. History of surgery in the past 28 days or with surgical wound not healed.
5. History of serious hemorrhage as defined by NCI CTCAE v5.0 grading.
6. Evidence of > grade 1 CNS hemorrhage on the baseline MRI scan.
7. History of recent hemoptysis.
8. Participants receiving therapeutic anticoagulation or antiplatelet therapy.
9. Participants with a history or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.
10. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease) requiring any treatment within the last 5 years.
11. History of organ transplant requiring immunosuppression.
12. History of active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
13. Prior use of anti-PD1 or PD-L1 immunotherapy or cellular therapy targeting PD-1/PD-L1 (or any NK cell therapy) for GBM.
14. Prior treatment with TTFields.
15. Uncontrolled seizures or neurological instability.
16. Should not require high-dose corticosteroids (eg, dexamethasone dose of ≤ 4 mg/day, or lowest dose to manage symptoms).
17. Other active malignancy requiring treatment.
18. Body weight ≤ 40 kg at screening.
19. Inadequate organ function, evidenced by the following laboratory results:

    1. ANC < 1,000 cells/mm3.
    2. Hemoglobin < 8 g/dL.
    3. Platelet count < 100,000 cells/mm3.
    4. Total bilirubin > 2 × ULN. For participants with documented Gilbert's syndrome, total bilirubin must be < 3 × ULN.
    5. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in participants with liver metastases).
    6. ALP levels > 2.5 × ULN (> 5 × ULN in participants with liver metastases, or > 10 × ULN in participants with bone metastases).
    7. Serum creatinine > 2.0 mg/dL or 177 µmol/L. Note: Each study site should use its institutional ULN to determine eligibility.
20. Clinically significant (ie, active) cardiovascular disease or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia. Participants with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
21. Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
22. Known hypersensitivity to any component of the study medication(s).
23. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol, including the use of the TTFields device as required or any psychiatric/social situation that would limit adherence to protocol.
24. Participation in an investigational drug study or receiving any investigational treatment within 28 days prior to study treatment or concurrent participation in any interventional clinical trial.
25. Pregnant and nursing women.
26. Active implanted medical device, a skull defect (such as, missing bone with no replacement) or bullet fragments. Examples of active electronic devices include deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators, and programmable shunts.
27. Known sensitivity to conductive hydrogels like the gel used on transcutaneous electrical nerve stimulation (TENS) electrodes.
28. A tumor located in the lower parts of the brain close to the spinal cord.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | From beginning of Cycle 1 (each cycle is 28 days) to 30 days after end of treatment study visit.
  TEAEs and SAEs graded using the NCI CTCAE v5.0
Incidence of clinically significant changes in comprehensive metabolic panel (CMP) | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and each subsequent treatment Cycle on Days 1 and Day 15 and at the end of treatment study visit.
  Standard blood chemistry panel made up of 14 separate chemistry measurements so can detect a range of abnormalities in blood sugar, nutrient balance, and liver and kidney health. Each clinical site will use their local laboratory upper limit of normal (ULN) range. The treating investigator will assess each result composing the CMP and determine if each result is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Hematology blood panel. | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and each subsequent treatment Cycle on Days 1 and Day 15 and at the end of treatment study visit.
  Blood test checking the levels for White Blood Cell, Red Blood Cell, Platelets, Hemoglobin, Hematocrit, Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils per unit volume. Each clinical site will use their local laboratory upper limit of normal (ULN) range. The treating investigator will assess each component of the Hematology panel and determine if each result is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Urinalysis. | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and each subsequent treatment Cycle on Days 1 and Day 15 and at the end of treatment study visit.
  Checking the appearance, concentration and content of urine for any abnormalities. Each clinical site will use their local laboratory upper normal limit (UNL) range. The treating investigator will assess each component of the urinalysis and determine if each result is within expected normal range or outside of the expected normal range.
12-lead Electrocardiogram (ECG) | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and each subsequent Cycle Day1 through to the end of treatment study visit.
  Perform 12-lead ECG as safety monitoring measurement. The parameters to be assessed for each one are the following: QT Interval, QTc Interval, QTcB Interval, QTcF Interval, PR Interval, QRS Duration and RR Interval with the unit in msec.
Incidence of clinically significant changes in Temperature | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and Cycle 2 on days 1, 2 and 15, followed by each subsequent treatment Cycle on Days 1 and 15 and on the end of treatment study visit.
  Temperature measured in either Fahrenheit or Celsius and for any abnormalities. Each site will assess to determine if temperature is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Heart Rate | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and Cycle 2 on days 1, 2 and 15, followed by each subsequent treatment Cycle on Days 1 and 15 and on the end of treatment study visit.
  Heart rate measured in beats/minute. Each site will assess to determine if heart rate is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Respiratory Rate | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and Cycle 2 on days 1, 2 and 15, followed by each subsequent treatment Cycle on Days 1 and 15 and on the end of treatment study visit.
  Respiratory rate measured in breaths/minute. Each site will assess to determine if respiratory rate is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Blood Pressure | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and Cycle 2 on days 1, 2 and 15, followed by each subsequent treatment Cycle on Days 1 and 15 and on the end of treatment study visit.
  Blood pressure measured in Systolic and Diastolic mmHg. Each site will assess to determine if blood pressure is within expected normal range or outside of the expected normal range.
Incidence of clinically significant changes in Oxygen Saturation | From baseline, pre-intervention, Cycle 1 (each cycle is 28 days) and Cycle 2 on days 1, 2 and 15, followed by each subsequent treatment Cycle on Days 1 and 15 and on the end of treatment study visit.
  A pulse oximeter measures oxygen saturation as a percentage. Determines the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin. Each site will assess to determine if oxygen saturation is within expected normal range or outside of the expected normal range.
Neurological assessment to grade Immune effector cell-associated neurotoxicity syndrome (ICANS) | On Cycle 1 (each cycle is 28 days) Day1, Day2, Day 15 and Day16, followed by each subsequent treatment Cycle on Days 1 and 15. Collection stops at the end of treatment study visit.
  Using a 10-point immune effector cell encephalopathy [ICE] score for the grading of ICANS. A score of 10 represents no impairment, 7-9 score is grade 1 ICANS, 3-6 score is grade 2 ICANS, 0-2 score is grade 3 ICANS and finally grade 4 ICANs is where cannot perform assessment of tasks.
Safety assessed by Cytokine Levels | From Cycle 1 (each cycle is 28 days) Day1, Day2, Day 15 and Day16, followed by each subsequent treatment Cycle on Day 1. Collection stops at the end of treatment study visit.
  The safety cytokine levels are TNF-α and IL-6

SECONDARY OUTCOMES:
Concentration of N-803 Pharmacokinetic (PK) | On Cycle 1 (each cycle is 28 days) and Cycle 3 on treatment days 1, 2, 3, 4, 5 and 8.
  Profile of each participant PK profile of N-803 from their serum sample
Concentration of PD-L1 t-haNK Pharmacokinetic (PK) | On Cycle 1 (each cycle is 28 days) and Cycle 3 on treatment days 1, 2, 3, 4, 5 and 8.
  Profile of each participant PK profile of PD-L1 t-haNK from their serum sample
Detection of Immunogenicity of N-803 | On Cycle 1 (each cycle is 28 days) Cycle 2 on treatment days 1 and 15, followed by Cycle 7 Day 1 and at the End of Treatment study visit.
  Detection of N-803 in each participant ADA serum blood samples
Detection of Immunogenicity of PD-L1 t-haNK | On Cycle 1 (each cycle is 28 days) Cycle 2 on treatment days 1 and 15, followed by Cycle 7 Day 1 and at the End of Treatment study visit.
  Detection of PD-L1 t-haNK in each participant ADA serum blood samples

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Chan Soon-Shiong Institute for Medicine (CSSIFM), El Segundo, California
  - Providence Medical Foundation, Fullerton, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No